CLINICAL TRIAL: NCT03888014
Title: Phase 4 Open Label Study Of Indocyanine Green Video Angiography (ICG-VA) And Comparative Utility Of Glow800 And FL800 Intraoperative ICG-VA Tools For Intracranial Lesions
Brief Title: Intraoperative Fluorescence With Augmented Reality
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00051776
Record Dates: First submitted 2019-02-22; First posted 2019-03-25 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Vascular; Lesion, Central Nervous System; Brain Tumor; Cerebral Aneurysm; Cerebral AVM
MeSH Terms: conditions — Brain Neoplasms; Intracranial Aneurysm; Intracranial Arteriovenous Malformations | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment group: The treatment group will consist of patients who require a medically necessary craniotomy. If an investigator deems that it will be useful to see blood vessels better with indocyanine green (ICG) videoangiography (VA), patients may be consented for the use if ICG VA using augmented reality (GLOW800). This will not add additional time or risk to their surgery
  Interventions: Device: GLOW800; Drug: indocyanine green (ICG)

INTERVENTIONS:
Device: GLOW800 — The treatment group will consist of patients who require a medically necessary craniotomy. If an investigator deems that it will be useful to see blood vessels better with indocyanine green (ICG) videoangiography (VA), patients may be consented for the use if ICG VA using augmented reality (GLOW800). This will not add additional time or risk to their surgery
Drug: indocyanine green (ICG) — This is a standard medication which can be given IV during a surgery to better visualize blood vessels under the microscope

SUMMARY:
This is a study looking at a new way to evaluate vascular problems or tumors in brain surgery patients using a standard & approved intravenous dye and augmented reality.

DETAILED DESCRIPTION:
This is a study investigating a new technique with an approved medication (ICG or indocyanine green) and using that and a near infrared mode on a standard operating room microscope to see the information provided for vascular or neoplastic (tumor related) neurosurgical problems. The technique uses the data from the microscope and using ICG with augmented reality overlaying the data into the microscope view (this is the new process). The technique is called GLOW800.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with a brain lesion requiring surgery and for whom ICG videoangiography would be used

Exclusion Criteria:

* allergy to ICG (indocyanine green)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with a brain lesion requiring surgery and for whom ICG videoangiography would be used
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Usefulness of Glow800 Technique | 48 hours
  Surgeon assessment of Glow800 compared to ICG-VA in usefulness

SECONDARY OUTCOMES:
Utility in Identifying a lesion | 48 hours
  Surgeon assessment of Glow800 vs ICG-VA in identifying vascular structures (useful, somewhat useful, not useful)
Surgical workflow | 48 hours
  Surgeon assessment of whether there is additional time (no additional time, <15 minutes additional time, <30 minutes additional time, >30 minutes additional time)
Additional Cost | 48 hours
  Surgeon assessment as to whether there is additional cost at surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States